CLINICAL TRIAL: NCT06854263
Title: ProspeCtive, muLti-site, Single-group, Open-lAbel Study to Evaluate the Safety and Performance of RADSAFE® Inks for radiaTion therapY Site Marking (CLARITY Study)
Brief Title: CLARITY Study - PMCF Study
Status: Not yet recruiting | Type: Observational
Sponsor: Laboratoires BIOTIC Phocea (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-RCB 2024-A01844-43
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Radiation Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mono-arm study
  Interventions: Device: skin marking for radiotherapy treatment

INTERVENTIONS:
Device: skin marking for radiotherapy treatment — skin marking for radiotherapy treatment

SUMMARY:
In the context of the Post-Market Clinical Follow-up (PMCF), this study aimed at evaluating the safety and performance of the RADSAFE® inks in the marking of the radiation field.

ELIGIBILITY:
Inclusion Criteria:

Male or female ≥18 years old, Cancer patient requiring radiotherapy, Patient requiring medical tattoo for treatment alignment, Intact skin at site of standard radiotherapy tattoos, ECOG performance status ≤2 (Karnofsky ≥60%), Able to provide written informed consent, Affiliated patient or beneficiary of a social security scheme.

Exclusion Criteria:

Previous medical tattoo of the targeted zone of treatment Known allergy to pigment ingredients, Infected or diseased skin, past or present, Affected organs close to the skin (eyes), Hypertrophic scars at site of radiotherapy tattoos, Carrying cardiac implant, Patient with blood clotting disorders, No consent to study participation, Under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision, An existing medical condition that, in the opinion of the Investigator, may put the subject at risk or compromise their participation in the study, Psychiatric illness/social situations that would limit compliance with study requirements, Females who are pregnant, lactating, or unwilling to use adequate birth control for the duration of the study, Personal objection to medical tattooing, Participation to another drug or medical device clinical interventional study that may interfere with the clinical investigation objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cancer requiring skin marking for radiotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of RADSAFE® for radiation therapy site skin-marking | From enrollment to the end of treatment at 8 weeks
  Rate of good or excellent skin marking visibility score (global evaluation) evaluated at the first session of radiotherapy delivery by two radiotherapy manipulators